CLINICAL TRIAL: NCT03032536
Title: A Randomized, Open-label, Multi-part Study of the Relative Oral Bioavailability of AL-3778 Tablets and Drug Interaction With Entecavir or Tenofovir Disoproxil Fumarate in Healthy Volunteers
Brief Title: Study of the Relative Oral Bioavailability of AL-3778 Tablets and Drug Interaction With Entecavir or Tenofovir Disoproxil Fumarate in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL-3778-1002; U1111-1187-4391 (Registry Identifier: WHO)
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis B; Chronic Hepatitis B; Viral Hepatitis B
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — NVR 3-778; entecavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Treatments A, B, C (Experimental): Part 1: Cross-Over
  * Treatment A: AL-3778 6 x 100-mg capsules (fasted) once.
  * Treatment B: AL-3778 2 x 300-mg tablets (fasted) once
  * Treatment C: AL-3778 2 x 300-mg tablets (high-fat meal) once.
  Interventions: Drug: AL-3778
- Treatments D, E, F (Experimental): Part 2 (optional): Cross-Over
  * Treatment D: AL-3778 2×300-mg tablets (fasted) once.
  * Treatment E: AL-3778 tablet Dose (fasted) once. Dose will match Treatment F dose and will be:
  * 1000mg: 2 x 500-mg OR
  * 800mg: 1 x 300-mg + 1 x 500-mg OR
  * 700mg: 1 x 200-mg + 1 x 500-mg
  * Treatment F: AL-3778 tablet Dose (high-fat meal) once. Dose will match Treatment E dose and will be:
  * 1000mg: 2 x 500-mg OR
  * 800mg: 1 x 300-mg + 1 x 500-mg OR
  * 700mg: 1 x 200-mg + 1 x 500-mg
  Interventions: Drug: AL-3778
- Treatment G (Experimental): Part 3: AL-3778 twice daily administered under fasted conditions for 14 days.
  Dose will be determined by Part 1 and/or Part 2 and will be one of the following tablet dosages:
  * 600mg: 2 x 300-mg OR
  * 1000mg: 2 x 500-mg OR
  * 800mg: 1 x 300-mg + 1 x 500-mg OR
  * 700mg: 1 x 200-mg + 1 x 500-mg
  Interventions: Drug: AL-3778
- Treatment H (Active Comparator): Part 3: Entecavir 0.5 mg once daily administered under fasted conditions for 14 days
  Interventions: Drug: Entecavir
- Treatment I (Experimental): Part 3: AL-3778 twice daily with entecavir 0.5 mg once daily both administered under fasted conditions for 14 days.
  AL-3778 dose will be determined by Part 1 and/or Part 2 and will be one of the following tablet dosages:
  * 600mg: 2 x 300-mg OR
  * 1000mg: 2 x 500-mg OR
  * 800mg: 1 x 300-mg + 1 x 500-mg OR
  * 700mg: 1 x 200-mg + 1 x 500-mg
  Interventions: Drug: AL-3778; Drug: Entecavir
- Treatment J (Active Comparator): Part 3: Tenofovir disoproxil fumarate 300 mg once daily administered under fasted conditions for 14 days
  Interventions: Drug: Tenofovir disoproxil fumarate
- Treatment K (Experimental): Part 3: AL-3778 twice daily and tenofovir disoproxil fumarate 300 mg once daily both administered under fasted conditions for 14 days.
  AL-3778 dose will be determined by Part 1 and/or Part 2 and will be one of the following tablet dosages:
  * 600mg: 2 x 300-mg OR
  * 1000mg: 2 x 500-mg OR
  * 800mg: 1 x 300-mg + 1 x 500-mg OR
  * 700mg: 1 x 200-mg + 1 x 500-mg
  Interventions: Drug: AL-3778; Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: AL-3778 — AL-3778 tablets or capsules
  Other Names: NVR 3-778, JNJ-63595948, ALS-003778
  Arms: Treatment G; Treatment I; Treatment K; Treatments A, B, C; Treatments D, E, F
Drug: Entecavir — Entecavir once daily for 14 days
  Arms: Treatment H; Treatment I
Drug: Tenofovir disoproxil fumarate — Tenofovir disoproxil fumarate once daily for 14 days
  Other Names: Viread
  Arms: Treatment J; Treatment K

SUMMARY:
This is an open-label, randomized, multi-part study to evaluate the relative oral bioavailability of a tablet formulation of AL-3778 (formerly NVR 3-778) administered under fasted and fed conditions (Parts 1 and 2) and the drug-drug interaction between AL-3778 and entecavir or tenofovir disoproxil fumarate (Part 3).

ELIGIBILITY:
Main Inclusion Criteria for All Subjects:

1. Subject has provided written consent.
2. In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and study restrictions and is likely to complete the study as planned.
3. Subject is in good health as deemed by the investigator, based on the totality of findings following a medical evaluation, including medical history, physical examination, laboratory tests and ECG.
4. Male or female, 18-60 years of age.
5. Body mass index 18-30 kg/m2, inclusive. The minimum weight is 50 kg.
6. A female subject is eligible to participate in this study if she is of non-childbearing potential (defined as females with a documented tubal ligation, bilateral oophorectomy or hysterectomy) or postmenopausal (defined as 12 months of spontaneous amenorrhea and follicle stimulating hormone level within the laboratory's reference range for postmenopausal females). A post-menopausal female receiving hormone replacement therapy who is willing to discontinue hormone therapy 28 days before study drug dosing and agrees to remain off hormone replacement therapy for the duration of the study may be eligible for study participation.
7. If male, subject is surgically sterile or practicing required forms of birth control until 6 months after the last dose of the study drug(s). Males must agree to refrain from sperm donation from check-in through 6 months after the last dose of the study drug(s).
8. Subject has been a nonsmoker and has not used nicotine or nicotine-containing products for at least 6 months.
9. Subjects who participated in Part 1 and/or Part 2 may participate in subsequent Part(s) upon satisfactory completion of a posttreatment visit, 7 days (+2 days) following the subject's last dose, and provided they continue to meet all of the inclusion criteria and none of the exclusion criteria.

Main exclusion criteria:

1. Subject is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 to 10 years.
2. Subject has a history of any illness that, in the opinion of the investigator, would confound the objectives or results of the study or poses an additional risk to the subject by their participation in the study.
3. Subject has an estimated creatinine clearance of ≤80 mL/min based on the Cockcroft-Gault equation; An actual creatinine clearance, as determined by a 24-hour urine collection, may be used in place of, or in conjunction with, the Cockcroft-Gault equation; subjects who have an actual or estimated creatinine clearance within 10% of 80 mL/min may be enrolled in the study at the discretion of the investigator.
4. Pregnant or nursing (lactating) females, confirmed by a positive human chorionic gonadotropin laboratory test or females contemplating pregnancy. Men whose female partners are pregnant or contemplating pregnancy from the date of screening until 6 months after their last dose of study drugs.
5. Clinically significant cardiovascular, respiratory, skeletal, renal, gastrointestinal, hematologic, hepatic, immunological, neurologic, endocrine, genitourinary abnormalities or disease or any other medical illness as determined by the investigator or Sponsor's Medical Monitor.
6. Subject has a history of malignancy except completely excised basal cell carcinoma or squamous cell carcinoma of the skin.
7. Subject lacks or has poor peripheral venous access.
8. Positive screening result for hepatitis B, hepatitis C and/or HIV serology.
9. Any condition that, in the opinion of the investigator, would compromise the study's objectives or the well-being of the subject or prevent the subject from meeting the study requirements.
10. Clinically significant abnormal ECG findings. Particularly, a history or family history of prolonged QT syndrome (eg, torsade de pointes) or sudden cardiac death.
11. ECG with PR >200 ms, QRS >120 ms, QTcF >450 ms, as assessed by triplicate 12-lead ECG at the screening visit.
12. Subject has had major surgery, or clinically significant blood loss or elective blood donation of significant volume (ie, >500 mL) within 60 days of first dose of study drug; >1 unit of plasma within 7 days of first dose of study drug.
13. Abnormal heart rate, respiratory rate, temperature or blood pressure values outside of the normal range (evaluated in a semi-recumbent or recumbent position after 5 minutes of rest). One repeat measurement after an additional 5 minutes of rest is permitted.
14. Evidence of active infection.
15. Unwilling to abstain from alcohol for at least 48 hours prior to the start of dosing through the study completion visit.
16. History of regular alcohol intake >7 units per week of alcohol for females and >14 units per week for males (one unit is defined as 10 g alcohol) within 3 months of the screening visit.
17. The subject has a positive screening or Day -1 drugs of abuse screen.
18. The use of concomitant medications, including prescription, over the counter medications, and herbal medications (such as St. John's Wort [Hypericum perforatum]) within 30 days prior to the first dose of study medication is excluded, unless approved by the Sponsor's Medical Monitor. Occasional use of ibuprofen/paracetamol/ acetaminophen is permitted.
19. Subject has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before the planned study drug.
20. Subject has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food.
21. Hypersensitivity to the active substances or to any of the excipients of AL-3778, entecavir or tenofovir disoproxil fumarate.
22. Subject has known allergy to heparin or history of heparin-induced thrombocytopenia.
23. Abnormal biochemistry or hematology laboratory results obtained at screening determined to be clinically significant by the Investigator. Screening ALT, AST, GGT, albumin, and total bilirubin must be within normal ranges. Creatine kinase >1.5 x ULN is exlusionary
24. Unwillingness or inability to comply with the study protocol for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
AL-3778, entecavir, tenofovir: Maximum observed plasma concentration (Cmax) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Area under the plasma concentration-time curve from time 0 to last measurable concentration (AUClast) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Area under the plasma concentration-time curve from time 0 to extrapolated to infinity (AUC∞) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Maximum observed plasma concentration on Day 1 (Cmax. Day 1) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1
AL-3778, entecavir, tenofovir: Minimum observed plasma concentration on Day 1 (Cmin, Day 1) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1
AL-3778, entecavir, tenofovir: Area under the plasma concentration-time curve from time 0 to dosing interval on Day 1 (AUC0-Τ, Day 1) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1
AL-3778, entecavir, tenofovir: Minimum observed plasma concentration (C_min) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22

SECONDARY OUTCOMES:
AL-3778, entecavir, tenofovir: Predose plasma concentrations (C_0-h) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Last observed plasma concentration (C_last) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Time of the maximum observed plasma concentration (T_max) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Time to last measurable plasma concentration (T_last) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Apparent oral clearance (CL/F) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Apparent volume of distribution (Vz/F) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Apparent terminal half-life (t½) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14 and once per day on Day 8, 10, 12, and 22
AL-3778, entecavir, tenofovir: Maximum observed plasma concentration on Day 14 (Cmax. Day 14) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 14
AL-3778, entecavir, tenofovir: Minimum observed plasma concentration on Day 14 (Cmin, Day 14) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 14
AL-3778, entecavir, tenofovir: Area under the plasma concentration-time curve from time 0 to dosing interval, tau, on Day 14 (AUC0-Τ, Day 14) | At 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours after dosing on Day 1 and 14
Incidence, nature, and severity of adverse events | Screening to Day 22
Changes in Vital Signs during and after study drug administration | Day 1 to Day 22
changes in physical examinations during and after study drug administration | Day 1 to Day 22
changes in clinical laboratory results during and after study drug administration | Day 1 to Day 22
changes in electrocardiogram results during and after study drug administration | Day 1 to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: William D Kennedy, MD, Study Director — Alios Biopharma Inc.
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Christchurch Clinical Studies Trust, Christchurch

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided per regulatory requirements.